CLINICAL TRIAL: NCT03966391
Title: Effectiveness of a Multi-faceted Knowledge Translation Intervention (The CARD System) for School Based Immunizations: a Cluster Trial
Brief Title: Effectiveness of CARD for Improving School-Based Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 036893
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Vaccination; Complications; Vaccine Adverse Reaction; Fear
Keywords: school vaccinations; pain management; knowledge translation; cluster trial
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Cluster trial involving 8 community health centres. They will be randomized to CARD or control (standard care) groups in a 1:1 ratio. Eligible schools (approximately 13/community health centre) will be included.
Who Masked: Participant
Masking Description: Students will not be aware of whether they are in the intervention or control group. Care providers who are trained in the intervention are aware of the group allocation. They will not communicate with care providers not trained in the intervention. Care providers that are trained in the intervention will not deliver care to participants in the control group and care providers that are not trained in the intervention will not deliver care to participants in the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARD (multi-faceted knowledge translation intervention) (Experimental): CARD will be integrated into the school vaccination program. This includes pre-vaccination day preparation (e.g., planning of clinic spaces, student and school staff education about CARD) and vaccination day activities (e.g., clinic set-up, processes for triaging students, implementing pain/ fear/fainting mitigation interventions from CARD during vaccination)
  Interventions: Other: Multi-faceted knowledge translation intervention
- Control (standard care) (No Intervention): There are no specific procedures being undertaken to plan or execute clinics. Usual practices will be instituted (i.e., no education specific to CARD, nor clinic set-up or execution to incorporate interventions for pain, fear or fainting)

INTERVENTIONS:
Other: Multi-faceted knowledge translation intervention — The intervention consists of education of relevant stakeholders of best practices and integration of best practices into the vaccination delivery program
  Other Names: CARD
  Arms: CARD (multi-faceted knowledge translation intervention)

SUMMARY:
Vaccination is estimated to have saved more lives in Canada than any other single intervention and is considered one of the most important advances in the prevention of disease. The process of vaccination, however, is stressful for individuals. School-based vaccinations in particular, are associated with high levels of fear and anxiety among students. This randomized cluster trial will implement a multi-faceted knowledge translation intervention called The CARD (C-Comfort A-Ask R-Relax D-Distract) System in school-based vaccinations and evaluate its effects on the experience of vaccination for students and implementation outcomes.

DETAILED DESCRIPTION:
The investigators developed a multi-faceted knowledge translation intervention called The CARD System to provide a framework for delivering vaccinations at school that integrates evidence-based strategies to mitigate pain, fear and fainting and promotes a student-centred approach to vaccination. CARD addresses 2 components of the vaccination delivery program: 1) pre-vaccination day preparation and 2) vaccination day activities. In a small controlled clinical trial in a public health unit in Niagara, Ontario, the investigators demonstrated benefits of CARD on student symptoms during vaccination, including fear, and dizziness-precursor of fainting, and satisfaction with CARD by all stakeholder groups (students, public health staff, school staff and parents). This study will evaluate CARD in a large cluster trial in Calgary, Alberta. This trial is the final phase of a 3-phase project, whereby the first 2 phases involve developing an implementation plan for the local context and evaluating feasibility of implementation.

Eight community health centres that provide vaccination services to schools in their regions will be randomized in a 1:1 ratio to CARD or control (usual practices). Data will be collected for vaccination services carried out in grade 6 and grade 9 students in participating schools for the academic year 2019-2020.

ELIGIBILITY:
Inclusion Criteria:

* grade 6 and 9 students eligible for vaccination at school
* public health staff in community health centre involved in the study
* school staff in a participating school involved in school vaccination
* parent of a student eligible for vaccination at school

Exclusion Criteria:

- unable to understand and read English

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8839 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Student fear | within 5 minutes after vaccination
  student self-reported fear during vaccination, rated on a 0-10 scale

SECONDARY OUTCOMES:
Student pain | within 5 minutes after vaccination
  student self-reported pain during vaccination, rated on a 0-10 scale
Student dizziness | within 5 minutes after vaccination
  student self-reported dizziness during vaccination, rated on a 0-10 scale
Student fainting | within 1 hour after vaccination
  student fainting during vaccination, yes/no, as assessed by immunizer
Student post-immunization stress-related responses | within 1 hour after vaccination
  student post-immunization stress-related responses, yes/no, as assessed by immunizer using the WHO Immunization Stress Responses Criteria
Utilization of coping strategies | within 5 minutes after vaccination
  use of individual coping strategies during vaccination (distraction, topical anesthetic, privacy, support person, deep breathing, muscle tension), yes/no, as assessed by immunizer using Documentation checklist
Uptake of vaccination | by end of school year
  proportion of students vaccinated (overall and for each vaccine)
Implementation success of CARD | within 3 months after vaccination clinics
  perceptions of implementation success of CARD program delivery as reported by CARD implementers (primary targets) using the CARD Global Impression Checklist, individual questions (5-point likert scale, higher number represents better outcome). This information will be supplemented with information from focus groups with implementers and study notes
Compliance with CARD | within 3 months after vaccination clinics
  percent compliance with CARD implementation as assessed by implementers using a CARD compliance checklist. This information will be supplemented with information from focus groups with implementers and study notes, as well as focus groups with other stakeholder groups (students, parents, school staff).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Alberta Health Services Public Health - Calgary Zone, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD